CLINICAL TRIAL: NCT02714153
Title: Bridge Occlusion Balloon Initial Use in Humans Study
Brief Title: Bridge Occlusion Balloon in Lead Extraction Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1602017220
Record Dates: First submitted 2016-03-04; First posted 2016-03-21 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: C.Surgical Procedure; Cardiac; Cardiac Dysrhythmia; Disorder of Pacing Function
Keywords: Lead extraction; Superior Vena Cava Tear; Pacemaker/Defibrillator lead extraction
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bridge Occlusion Balloon (Experimental): Bridge Balloon catheter is designed to be used for temporary vessel occlusion of the superior vena cava in applications including perioperative occlusion and emergency control of hemorrhage associated with vascular tears that may occur during lead extraction procedures.
  Interventions: Device: Bridge Balloon

INTERVENTIONS:
Device: Bridge Balloon — The Bridge Balloon will be used in a non-emergent setting to allow for evaluation of how best to integrate this new technology into the investigators clinical practice. The study will focus on the effect of the Bridge balloon on the patient preparation clinical workflow, ease of insertion/positioning/deployment, and the ability to recognize proper inflation and vein sealing under fluoroscopy.
  Other Names: Bridge Occlusion Balloon, Spectranetics

SUMMARY:
To evaluate the use of an occlusion balloon (Bridge™ Occlusion Balloon, Spectranetics) within the Superior Vena Cava in lead extraction patients.

DETAILED DESCRIPTION:
This study will evaluate the use of an occlusion balloon (Bridge™ Occlusion Balloon, Spectranetics) within the Superior Vena Cava in lead extraction patients. This will be performed in a non-emergent setting to allow for evaluation of how best to integrate this new technology into the investigators clinical practice. The study will focus on the effect of the Bridge balloon on the patient preparation clinical workflow, ease of insertion/positioning/deployment, and the ability to recognize proper inflation and vein sealing under fluoroscopy. Understanding these factors will help build a more robust clinical workflow with the goal of better patient outcomes in the case of an Superior Vena Cava injury. The images and data generated during this study can help in dissemination of the practical use knowledge to fellow lead extractors.

At the time of the protocol registration, the timeframe 12 months was entered, this was actually the anticipated length of the study at registration. The timeframe was corrected to 33 minutes (average time) at the time of results entry.

ELIGIBILITY:
Inclusion Criteria:

* Subject age more than 18 years
* Lead extraction patients

Exclusion Criteria:

Lead extraction patients with:

* Superior Vena Cava occlusion or stenosis.
* Significant vegetation.
* Hemodynamic instability.
* Class IV heart failure
* Creatinine > 2.0mg/dL
* Patients > 85 years old

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04; Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jude Clancy, MD, Principal Investigator — Yale University
Locations (7):
- United States (7):
  - University of Miami Hospital, Miami, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - United Hospital, Saint Paul, Minnesota
  - Cooper University Health Care, Camden, New Jersey
  - Sanger Heart & Vascular Institute Carolinas HealthCare System, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bridge Occlusion Balloon
Started | 23
Completed | 22
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bridge Occlusion Balloon
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23
Comorbidities [Count of Participants; unit: Participants]
  Congenital Heart Disease | 1
  Diabetes Mellitus | 6
  Coronary Artery Disease | 11
New York Heart Association Class [Count of Participants; unit: Participants] — NYHA Classification - The Stages of Heart Failure: Class I - No symptoms; Class II - Mild symptoms; Class III - Marked limitation in activity due to symptoms; Class IV - Severe limitations.
  Participants
    I | 2
    II | 5
    III | 13
    IV | 3
Ejection Fraction [Mean (Standard Deviation); unit: percent] — Ejection fraction (EF) is a measurement, expressed as a percentage, of how much blood the left ventricle pumps out with each contraction.
  percent | 43 (15)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.05 (0.29)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Balloon Occlusion of Superior Vena Cava
Description: After Bridge Balloon deployment and inflation, the degree of blood vessel occlusion will be reported. Measurements will be calculated from fluoroscopic images (using x-ray machine) and venograms (images with injection of contrast agent). Successful balloon occlusion of the superior vena cava (SVC) is defined as >90% occlusion of the SVC by visual estimate using conventional venography.
Time Frame: 33 minutes (average time)
Population: All patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Occlusion Balloon
Number analyzed (Participants) | 23
Participants
  First Balloon Deployment | 18
  Reposition and Reinflation | 5

2. Secondary Outcome: Time of Bridge Balloon Deployment
Description: Time will be calculated in seconds starting from opening the Bridge Balloon Package up to full balloon deployment.
Time Frame: 33 minutes (average time)
Population: All patients.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Bridge Occlusion Balloon
Number analyzed (Participants) | 23
seconds | 121 (50)

3. Secondary Outcome: Number of Participants With Changes in Heart Rate at One Year
Description: Heart Rate (in beat per minute) will be collected at 5 points: baseline, after guidewire insertion, at the time of balloon inflation, immediately post deflation and 5 minutes post deflation (all during the procedure itself). This outcome will be reported at the end of the study as if there were any unacceptable or no unacceptable changes in the hemodynamics over the course of the 12 month period.
Time Frame: 1 year
Population: All patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Occlusion Balloon
Number analyzed (Participants) | 23
Participants
  Unacceptable Changes | 0
  No Unacceptable Changes | 23

4. Secondary Outcome: Number of Participants With Changes in Blood Pressure at One Year
Description: Blood pressure in mmHg will be collected at 5 points: baseline, after guidewire insertion, at the time of balloon inflation, immediately post deflation and 5 minutes post deflation (all during the procedure itself). This outcome will be reported at the end of the study as as if there were any unacceptable or no unacceptable changes in the hemodynamics over the course of the 12 month period..
Time Frame: 1 year
Population: All patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Occlusion Balloon
Number analyzed (Participants) | 23
Participants
  Unacceptable Changes | 0
  No Unacceptable Changes | 23

5. Secondary Outcome: Number of Participants With Changes in SPO2 at One Year
Description: SPO2 will be collected at 5 points: baseline, after guidewire insertion, at the time of balloon inflation, immediately post deflation and 5 minutes post deflation (all during the procedure itself). This outcome will be reported at the end of the study as if there were any unacceptable or no unacceptable changes in the hemodynamics over the course of the 12 month period..
Time Frame: 1 year
Population: All patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Occlusion Balloon
Number analyzed (Participants) | 23
Participants
  Unacceptable Changes | 0
  No Unacceptable Changes | 23

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Bridge Occlusion Balloon
All-Cause Mortality (participants affected / at risk) | 1/23
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bridge Occlusion Balloon (N=23)
SVC Tear (Vascular disorders) | 1 (1) — An SVC tear occurred intraoperatively during the course of the study. The procedure was thoroughly reviewed by the data safety monitoring committee and it was concluded deployment of the balloon had no relation to the adverse outcome of the SVC tear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT02714153/Prot_001.pdf
  • Statistical Analysis Plan (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT02714153/SAP_000.pdf